CLINICAL TRIAL: NCT06333743
Title: Efficacy, Acceptability, and Safety of Laser Ablation in the Treatment of High-grade Cervical Lesions: a Randomized Clinical Trial
Brief Title: Laser Ablation in the Treatment of High-grade Cervical Lesions
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Obstetrics & Gynecology Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZhuLan
Record Dates: First submitted 2024-02-25; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: High-Grade Squamous Intraepithelial Lesions
Keywords: HSIL; laser ablation
MeSH Terms: conditions — Squamous Intraepithelial Lesions | interventions — Laser Therapy; Conization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laser ablation treatment (Experimental): Laser vaporization is performed using a carbon dioxide laser under colposcopy. All patients received 1% mepivacaine hydrochloride paracervix block. No general anesthesia was used. Before laser vaporization began, scaly columnar nodules were visible in all patients. The evaporation depth is 8-10mm, and the edge is 5mm from the abnormal discovery or transition area.
  Interventions: Procedure: laser ablation
- LEEP or conization treatment (Active Comparator): The cervix was stained with iodine solution and the diseased lesion was visualized. LEEP or conization was performed to a depth of approximately 1.5 cm to resect disease in the cervical canal.
  Interventions: Procedure: LEEP or Conization

INTERVENTIONS:
Procedure: laser ablation — Research has confirmed that laser ablation treatment of cervical HSIL is effective and feasible.
  Arms: laser ablation treatment
Procedure: LEEP or Conization — The most common treatment for HSIL is LEEP or conization of the cervical lesion, but there are several perinatal complications involved in this surgery.
  Arms: LEEP or conization treatment

SUMMARY:
Cervical laser ablation is an effective, minimally invasive treatment with a low incidence of perinatal complications and minimal impact on fertility. Research has confirmed that laser ablation treatment of cervical HSIL (including CIN2 and CIN3) is effective and feasible and is useful for young CIN3 patients who wish to get pregnant in the future. There have been no randomized clinical trials of laser ablation therapy for cervical HSIL in Chinese women. This study focuses on the application of laser ablation in the treatment of cervical HSIL, explores the efficacy, feasibility, and safety of laser ablation in the treatment of cervical HSIL, and strives to promote the reasonable application of laser ablation in the treatment of cervical HSIL.

DETAILED DESCRIPTION:
1. Background This study focuses on the application of laser ablation in the treatment of cervical HSIL, explores the efficacy, feasibility, and safety of laser ablation in the treatment of cervical HSIL, and strives to promote the reasonable application of laser ablation in the treatment of cervical HSIL.
2. Research objects Young patients with cervical HSIL underwent colposcopic evaluation, completed cervical biopsy, and were pathologically confirmed to be eligible for ablation.
3. Methods 3.1 Sample size This study was a randomized controlled trial with parallel design. HSIL recurrence rate was the primary endpoint. According to previous literature reports, it is estimated that the recurrence rate of HSIL in the laser treatment group is 15%. The recurrence rate of HSIL in the resection group was 5%. Let α=0.05 (both sides), hold =0.80. Using PASS 11 software, the sample size of both groups was 138 cases. Assuming that the loss of follow-up rate of the study subjects was 10%, the sample size of each group was 138÷0.9=154 cases. Therefore, 308 patients were intended to be included in the study.

   3.2 Statistical methods SPSS 24.0 software will be used for statistical analysis of all data. Measurement data with normal distribution will be described by mean ± standard deviation. Independent sample t-test or rank sum test will be used for inter-group comparison, and paired sample t-test will be used for intra-group comparison before and after treatment. Counting data will be expressed as examples or percentages (%), and the Chi-square test will be used for comparison between groups. The Kaplan-Meier method will be used to calculate the recurrence rate, and the rank sum test will be used to evaluate the difference between the two groups. Cox regression model will be used to analyze the factors influencing prognosis. P < 0.05 will be considered statistically significant.
4. Results The primary endpoint is the HSIL recurrence rate at 12 months after treatment.

Other subjects were secondary study endpoints shown as follows:

Intraoperative and postoperative complications and side effects, including bleeding, pain, infection, cervical secretions, and healing; Psychological state change; Satisfaction; Cervical length; Recurrence rate; Fees

ELIGIBILITY:
Inclusion Criteria:

1. < 40-year-old
2. Cervical HSIL confirmed by colposcopic biopsy pathology
3. Cervical transformation zone type 1 or 2
4. The lesion is completely visible and does not extend into the cervical canal, and the lesion area is less than 50% of the cervical surface area
5. Colposcopic evaluation ruled out invasive cancer
6. Voluntary participation in the study with full and informed consent

Exclusion Criteria:

1. Cervical transformation zone type 3
2. Glandular epithelial lesions
3. Lesions greater than 50% of cervical surface area, or with vaginal and vulvar intraepithelial lesions
4. The upper margin of the lesion was not visible or extended into the cervical canal
5. Cervical tube sampling was diagnosed with CIN2+ or CIN that could not be graded
6. Cervical biopsy is not sufficient to confirm a tissue diagnosis
7. Suspected invasive cancer
8. History of cervical surgery
9. Pregnancy or planning a pregnancy during study participation
10. Autoimmune or immune deficiency diseases
11. Long-term use of immunosuppressive drugs

Max Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 308 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
the rate of HSIL recurrence | 12 months after treatment
  12 months after the treatment, TCT, HPV, colposcopy, and biopsy will be tested again. If the result of the biopsy is HSIL again, we will record it as HSIL recurrence.

SECONDARY OUTCOMES:
the satisfaction with the treatment | 8 weeks and 12 months after treatment
  after the treatment, patients will fill in a questionnaire to describe their degree of satisfaction with the treatment
the length of the cervix | 8 weeks and 12 months after treatment
  the length of the cervix will be measured by B-ultrasound
Psychological state change related to the treatment | 8 weeks and 12 months after treatment
  State-Trait Anxiety Inventory，STAI-Form Y will be used to measure the patients' psychological state after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Lan Zhu, MD, Principal Investigator — Peking Union Medical College Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Perkins RB, Guido RS, Castle PE, Chelmow D, Einstein MH, Garcia F, Huh WK, Kim JJ, Moscicki AB, Nayar R, Saraiya M, Sawaya GF, Wentzensen N, Schiffman M; 2019 ASCCP Risk-Based Management Consensus Guidelines Committee. 2019 ASCCP Risk-Based Management Consensus Guidelines for Abnormal Cervical Cancer Screening Tests and Cancer Precursors. J Low Genit Tract Dis. 2020 Apr;24(2):102-131. doi: 10.1097/LGT.0000000000000525. No abstract available. PMID 32243307
- [Background] Sadler L, Saftlas A, Wang W, Exeter M, Whittaker J, McCowan L. Treatment for cervical intraepithelial neoplasia and risk of preterm delivery. JAMA. 2004 May 5;291(17):2100-6. doi: 10.1001/jama.291.17.2100. PMID 15126438
- [Background] Kyrgiou M, Koliopoulos G, Martin-Hirsch P, Arbyn M, Prendiville W, Paraskevaidis E. Obstetric outcomes after conservative treatment for intraepithelial or early invasive cervical lesions: systematic review and meta-analysis. Lancet. 2006 Feb 11;367(9509):489-98. doi: 10.1016/S0140-6736(06)68181-6. PMID 16473126
- [Background] Fallani MG, Penna C, Fambrini M, Marchionni M. Laser CO2 vaporization for high-grade cervical intraepithelial neoplasia: a long-term follow-up series. Gynecol Oncol. 2003 Oct;91(1):130-3. doi: 10.1016/s0090-8258(03)00440-2. PMID 14529672
- [Result] Mariya T, Nishikawa A, Sogawa K, Suzuki R, Saito M, Kawamata A, Shimizu A, Nihei T, Sonoda T, Saito T. Virological and cytological clearance in laser vaporization and conization for cervical intra-epithelial neoplasia grade 3. J Obstet Gynaecol Res. 2016 Dec;42(12):1808-1813. doi: 10.1111/jog.13113. Epub 2016 Aug 16. PMID 27526956
- [Result] Zhang L, Sauvaget C, Mosquera I, Basu P. Efficacy, acceptability and safety of ablative versus excisional procedure in the treatment of histologically confirmed CIN2/3: A systematic review. BJOG. 2023 Jan;130(2):153-161. doi: 10.1111/1471-0528.17251. Epub 2022 Jul 4. PMID 35689493
- [Result] Yoon BS, Seong SJ, Song T, Kim ML, Kim MK. Risk factors for treatment failure of CO2 laser vaporization in cervical intraepithelial neoplasia 2. Arch Gynecol Obstet. 2014 Jul;290(1):115-9. doi: 10.1007/s00404-014-3148-1. Epub 2014 Jan 24. PMID 24458427
- [Result] Kodama K, Yahata H, Okugawa K, Tomonobe H, Yasutake N, Yoshida S, Yagi H, Yasunaga M, Ohgami T, Onoyama I, Asanoma K, Hori E, Shimokawa M, Kato K. Prognostic outcomes and risk factors for recurrence after laser vaporization for cervical intraepithelial neoplasia: a single-center retrospective study. Int J Clin Oncol. 2021 Apr;26(4):770-776. doi: 10.1007/s10147-020-01848-x. Epub 2021 Jan 4. PMID 33394202
- [Result] Inaba K, Nagasaka K, Kawana K, Arimoto T, Matsumoto Y, Tsuruga T, Mori-Uchino M, Miura S, Sone K, Oda K, Nakagawa S, Yano T, Kozuma S, Fujii T. High-risk human papillomavirus correlates with recurrence after laser ablation for treatment of patients with cervical intraepithelial neoplasia 3: a long-term follow-up retrospective study. J Obstet Gynaecol Res. 2014 Feb;40(2):554-60. doi: 10.1111/jog.12196. Epub 2013 Oct 11. PMID 24118526
- See also: WHO guidelines for the use of thermal ablation for cervical pre-cancer lesions — http://www.ncbi.nlm.nih.gov/books/NBK549182/